CLINICAL TRIAL: NCT02560025
Title: A Phase II Study of the Aurora A Kinase Inhibitor Alisertib in Combination With 7+3 Induction Chemotherapy in Patients With High-risk Acute Myeloid Leukemia
Brief Title: Phase II Trial of Alisertib With Induction Chemotherapy in High-risk AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-334
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — MLN 8237; Cytarabine; Idarubicin; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alisertib / MLN8237 (Experimental): Participants will initially receive 7+3 induction chemotherapy, consisting of cytarabine and concurrent idarubicin (or daunorubicin if appropriate). Oral alisertib, at 30mg twice daily, will begin on day 8, and will continue for 7 days. During induction, patients with residual disease at day 14 may have re-induction with "5+2" chemotherapy, but will not receive additional dosing of alisertib at that time. Following count recovery after induction, if patients proceed to consolidative cycles of therapy with cytarabine, they will receive alisertib at day 6 following conclusion of cytarabine administration. Upon count recovery following consolidation, alisertib will be resumed for 7 days, followed by 14 days off, and will be continued as 21-day cycles of maintenance, for up to 12 cycles.
  Interventions: Drug: Alisertib; Drug: Cytarabine; Drug: Idarubicin; Drug: Daunorubicin

INTERVENTIONS:
Drug: Alisertib
  Other Names: MLN8237
Drug: Cytarabine
  Other Names: Cytosine Arabinoside
Drug: Idarubicin
  Other Names: Idarubicin hydrochloride
Drug: Daunorubicin — Can be used in place of idarubicin
  Other Names: Cerubidine®

SUMMARY:
This research study is studying a targeted therapy (a form of treatment that uses drugs or other substances to identify and attack specific types of cancer cells with less harm to normal cells) as a possible treatment for high-risk acute myeloid leukemia.

The names of the study interventions involved in this study are:

* Alisertib / MLN8237
* Cytarabine / Cytosine Arabinoside
* Idarubicin / Idarubicin hydrochloride
* Daunorubicin (Can be used in place of idarubicin)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

As part of this research study, the participant will take alisertib in combination with conventional chemotherapies, idarubicin and cytarabine. Alisertib has not been approved by the FDA (U.S. Food and Drug Administration) for acute myeloid leukemia (AML). However, cytarabine and idarubicin have both been approved by the FDA for treatment of AML. It also means that the FDA (U.S. Food and Drug Administration) has not approved giving alisertib with idarubicin and cytarabine for use in participants, including participants with this type of cancer.

Earlier pre-clinical studies and clinical trials have suggested the alisertib may have clinical promise as a single agent in acute myeloid leukemia. Alisertib is a selective small molecule inhibitor of Aurora A kinase, an enzyme which may play a role in the survival of leukemia cells. Alisertib is being studied for the treatment of advanced malignancies, including AML. Essentially, this means that alisertib may work to halt the growth of malignancy (abnormal cells dividing without control and invading nearby tissues) through a targeted mechanism. By combining alisertib with standard chemotherapy, the hope is to enhance the efficacy of current treatment used for acute myeloid leukemia. An earlier study of this combination has completed accrual, and demonstrated that the regimen is well tolerated.

Through this study, the investigators would like to determine if the addition of alisertib to standard 7+3 chemotherapy improves efficacy as measured by the rate of complete remission (a decreased or disappearance of signs and symptoms of cancer).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed, newly diagnosed high-risk acute myeloid leukemia, as defined by at least one of the following criteria

  * Age greater than or equal to 65 years
  * Poor risk karyotype, as per Leukemianet criteria
  * Antecedent or underlying myelodysplastic syndrome or myeloproliferative neoplasm
  * AML with MDS-related changes
* Adults, age 18 years or older at the time of diagnosis, eligible for standard induction chemotherapy according to their treating physician.
* ECOG performance status 0-2 (Karnofsky ≥60%, see Appendix A)
* Left ventricular ejection fraction > 50% as measured by echocardiogram or MUGA scan
* Must not have received systemic antineoplastic therapy including radiation therapy within 14 days of the study enrollment, except hydroxyurea or 6-mercaptopurine for the purposes of cytoreduction. Patients may also have received all-trans retinoic acid (ATRA) if there is an early suspicion of acute promyelocytic leukemia (APL, M3-AML), although if confirmed to have APL these patients will be excluded from the study.
* Adequate renal function as defined by: calculated creatinine clearance ≥40 mL/min (Cockcroft-Gualt Formula)
* Direct bilirubin < 2.0 x upper limit of normal (ULN), SGOT (AST) and SGPT (ALT)< 2.5 x ULN. AST and/or ALT may be up to 5X ULN if thought to be secondary to leukemia.
* The effects of alisertib on the developing human fetus are unknown. For this reason and because other chemotherapeutic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and 6 months after completion of therapy.
* Subject must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after alisertib administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients will be excluded from this study if they do not otherwise fulfill criteria mentioned in bullet 3.1.1, and are found to harbor "intermediate" or "favorable" risk cytogenetics 41:
* In such patients, a sample to evaluate patient cytogenetics will be sent at the time of diagnosis per standard clinical care and the absence of favorable or intermediate-risk cytogenetics must be confirmed by Day 8. If the cytogenetic analysis reveals that the patient harbors non-poor risk cytogenetics, or if the cytogenetic results are not received prior to Day 8, the participant will be removed from the study.
* Patients with acute bilineal/biphenotypic leukemia
* Participants who have had chemotherapy or radiotherapy within 14 days prior to entering the study, except for hydroxyurea or 6-MP as noted.
* Participants who are receiving or have received any other investigational agents within 14 days of enrollment.
* Chemo-, hormono-, radio- or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug
* Persistence of clinically relevant therapy related toxicity from previous anti-cancer therapy
* Prior allogeneic bone marrow or organ transplantation
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Current clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukemic CNS involvement (no lumbar puncture required, clinical assessment per investigator's judgment is sufficient).
* If applicable, patient with ≥Grade 2 peripheral neuropathy within 14 days before enrollment
* Prior treatment with alisertib
* Known history of hepatitis C infection or suspected currently active hepatitis C infection. Known or suspected history of hepatitis B infection will be excluded when any of the following conditions are met:

  * Received hematopoietic stem cell transplantation (either allogenic or autologous), or
  * Received any rituximab-containing treatment regimen in the last 12 months before entering the study, or
  * Tested positive for the presence of at least 1 of the following 3 markers in blood (evaluated at screening): hepatitis B surface antigen (HBsAG), antibodies against hepatitis B core antigen (anti-HBc), or hepatitis B viral load (HBV DNA).
* Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF <50%, as measured by MUGA scan or echocardiogram). Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Known hypersensitivity to the trial drugs or other contraindication to standard "7+3" induction chemotherapy.
* Known history of uncontrolled sleep apnea syndrome, or sleep apnea requiring supplemental oxygen, and other conditions that could result in excessive daytime sleepiness.
* A medical condition requiring use of proton pump inhibitors (PPIs); or histamine 2 (H2) receptor antagonists. Patients who intermittently use these medications, must meet the following criteria:

  * No use of PPIs within 5 days before the first dose of alisertib
  * No use of H2 antagonist or pancreatic enzymes within 24 hours before the first dose of alisertib
* Patients with mental deficits or psychiatric conditions that preclude them from giving informed consent or following protocol.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known GI disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib. Examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease.
* Pregnant women are excluded from this study because alisertib, along with standard induction chemotherapy, carries the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with alisertib as well as cytarabine and idarubicin, breastfeeding should be avoided. Confirmation that the subject is not pregnant must be established by a negative serum ß-human chorionic gonadotropin ( ß-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Although not absolute exclusion criteria, because of known drug-drug interactions, below are issues that should be considered during enrollment:
* Treatment with clinically significant enzyme-inducing drugs, including known P-glycoprotein inducers (including St John's wort and rifampicin) should be used only if absolutely necessary and considered to be the best available choice for the patient. If possible, it is recommended that alternatives to known substrates, inhibitors or inducers of P-glycoprotein be considered. Cases should be discussed with the principal investigator, and may be allowed as per his/her discretion.

  * Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
  * Patients who are otherwise felt unable to comply with the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brunner AM, Blonquist TM, DeAngelo DJ, McMasters M, Fell G, Hermance NM, Winer ES, Lindsley RC, Hobbs GS, Amrein PC, Hock HR, Steensma DP, Garcia JS, Luskin MR, Stone RM, Ballen KK, Rosenblatt J, Avigan D, Nahas MR, Mendez LM, McAfee SL, Moran JA, Bergeron M, Foster J, Bertoli C, Manning AL, McGregor KL, Fishman KM, Kuo FC, Baltay MT, Macrae M, Burke M, Behnan T, Wey MC, Som TT, Ramos AY, Rae J, Lombardi Story J, Nelson N, Logan E, Connolly C, Neuberg DS, Chen YB, Graubert TA, Fathi AT. Alisertib plus induction chemotherapy in previously untreated patients with high-risk, acute myeloid leukaemia: a single-arm, phase 2 trial. Lancet Haematol. 2020 Feb;7(2):e122-e133. doi: 10.1016/S2352-3026(19)30203-0. Epub 2019 Dec 11. PMID 31837959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alisertib / MLN8237
Started | 42
Completed | 39
Not Completed | 3
Not completed — Ineligible after consent/ registration | 3

BASELINE CHARACTERISTICS:
Population: The three participants found to be ineligible after enrollment were excluded from the analysis
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 67 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39
Cytogenetic Risk [Count of Participants; unit: Participants] — Higher risk represents an increased chance that the participant will experience undesirable disease outcomes.
  Participants
    High | 13
    Intermediate | 26
Median White Blood Cell (WBC) Count [Median (Full Range); unit: Thousand WBC/ microliter blood] | 3.2 [0.4 to 59.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved Complete Remission
Description: The number of participants that achieved a best overall response of complete remission while on study.
  Complete remission (CR): Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/μL and a platelet count of 100,000/μL, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, existing extramedullary disease. If possible, at least one bone marrow biopsy should be performed to confirm CR.
Time Frame: From the start of treatment until the end of study treatment, up to approximately 10 months
Population: The three participants found to be ineligible after enrollment were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 39
Participants | 20

2. Primary Outcome: Number of Participants That Achieved Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: The number of participants that achieved a best overall response of CRi while on study.
  Complete Remission with Incomplete Blood Count Recovery (CRi): Same as for CR but without achievement of ANC at least 1000/uL (CRi) and/or platelet count of 100,000/uL (CRp).
Time Frame: From the start of treatment until the end of study treatment, up to approximately 10 months
Population: The three participants found to be ineligible after enrollment were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 39
Participants | 5

3. Secondary Outcome: 1 Year Overall Survival Rate
Description: The percentage of participants alive at one year
Time Frame: 1 Year
Population: The three participants found to be ineligible after enrollment were excluded from the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 39
percentage of participants | 50 [34 to 66]

4. Secondary Outcome: Median Relapse Free Survival
Description: The median amount of time from achieving a complete remission to the first of disease recurrence or death. RFS applies only to the subset of patients who achieve a CR+CRi at the end of induction therapy.
  * Complete remission (CR): Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/μL and a platelet count of 100,000/μL, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, existing extramedullary disease. If possible, at least one bone marrow biopsy should be performed to confirm CR.
  * Complete remission with incomplete blood count recovery (CRi): Same as CR but without achievement of specified ANC and/or platelet count
  * Recurrence/ morphologic relapse: reappearance of leukemic blasts in the peripheral blood or >5% blasts in the bone marrow not attributable to any other cause
Time Frame: From the time of treatment response until death or disease progression (up to about one year)
Population: Participants that achieved a complete response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 20
Months | NA [7.1 to NA] — The median value and the upper limit of the confidence interval are not defined due to an insufficient number of patients experiencing relapse

5. Secondary Outcome: Median Duration of Remission
Description: The median amount of time from first achieving remission to disease progression (with patients censored at death).
  * Complete remission (CR): Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/μL and a platelet count of 100,000/μL, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, existing extramedullary disease. If possible, at least one bone marrow biopsy should be performed to confirm CR.
  * Complete remission with incomplete blood count recovery (CRi): Same as CR but without achievement of specified ANC and/or platelet count
  * Recurrence/ morphologic relapse: reappearance of leukemic blasts in the peripheral blood or >5% blasts in the bone marrow not attributable to any other cause
Time Frame: From the time of first remission to disease progression or death, median duration of 12.8 months
Population: Participants that achieved a complete response
Measure: Median (Full Range); unit: Months
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 20
Months | 12.8 [11.5 to 14.7]

6. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4). Adverse events were considered to be Serious Adverse Events (SAE) if they were grade 3 or greater and deemed to be possibly, probably, or definitely related to the study treatment.
Time Frame: From the start of treatment until 30 days after the last dose of a study drug is received, up to approximately 11 months
Population: The three participants found to be ineligible after enrollment were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib / MLN8237
Number analyzed (Participants) | 39
Participants | 27

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the last dose of a study drug is received, up to approximately 11 months
Description: The adverse events reported in the serious adverse event section represent CTCAE 4 grade 3 or greater adverse events that were deemed to be possibly, probably, or definitely related to study treatment.
Arm/Group | Alisertib / MLN8237
All-Cause Mortality (participants affected / at risk) | 20/39
Serious Adverse Events (participants affected / at risk) | 27/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib / MLN8237 (N=39)
Alanine aminotransferase increased (Investigations) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 3 (4)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 12 (14)
Platelet count decreased (Investigations) | 12 (17)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib / MLN8237 (N=39)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Acute kidney injury (Renal and urinary disorders) | 5 (8)
Alanine aminotransferase increased (Investigations) | 12 (14)
Alkaline phosphatase increased (Investigations) | 15 (20)
Anal fistula (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 13 (25)
Anorexia (Metabolism and nutrition disorders) | 23 (28)
Anxiety (Psychiatric disorders) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 10 (13)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Blood bilirubin increased (Investigations) | 13 (18)
Blurred vision (Eye disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3)
Catheter related infection (Infections and infestations) | 2 (2)
Chills (General disorders) | 7 (7)
Colitis (Gastrointestinal disorders) | 5 (5)
Confusion (Psychiatric disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Creatinine increased (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Delirium (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 29 (35)
Dizziness (Nervous system disorders) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Edema limbs (General disorders) | 7 (7)
Enterocolitis (Gastrointestinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 22 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (20)
Fever (General disorders) | 11 (14)
Floaters (Eye disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders - Other, Lack of Appetite (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (10)
Hematoma (Vascular disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5)
Hypertension (Vascular disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Hypotension (Vascular disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Insomnia (Psychiatric disorders) | 9 (9)
Localized edema (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 10 (10)
Mucositis oral (Gastrointestinal disorders) | 15 (17)
Nausea (Gastrointestinal disorders) | 21 (27)
Neutrophil count decreased (Investigations) | 9 (15)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Platelet count decreased (Investigations) | 11 (31)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (18)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sepsis (Infections and infestations) | 6 (7)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus pain (Nervous system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Syncope (Nervous system disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 4 (4)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (9)
White blood cell decreased (Investigations) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT02560025/Prot_SAP_000.pdf